CLINICAL TRIAL: NCT04990167
Title: Tiotropium vs. Inhaled Corticosteroids in Children With Nonatopic Asthma Pilot Study
Brief Title: Tiotropium vs. Inhaled Corticosteroids in Children With Nonatopic Asthma Pilot Study (TioNAAP)
Acronym: TioNAAP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult enrollment
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Gerardo Vazquez Garcia, Faculty Physician, Nemours Children's Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1753113-1
Record Dates: First submitted 2021-06-17; First posted 2021-08-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Asthma in Children
Keywords: Nonatopic
MeSH Terms: interventions — Tiotropium Bromide

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, open-label crossover pilot feasibility trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tiotropium arm (Experimental): Subjects on this arm will start the study on tiotropium for 6 weeks. Received prescribed asthma controller medication for 2 weeks " washout" and complete 6 week on the prescribed asthma controller medication.
  Interventions: Drug: Tiotropium Bromide
- ICS arm (Active Comparator): Subjects on this arm will start the study on the prescribed asthma medication for 6 weeks. Received prescribed asthma controller medication for 2 weeks " washout" and complete 6 week on Tiotropium.
  Interventions: Drug: Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium Bromide — Using Tiotropium as a single agent asthma controller medication

SUMMARY:
Most children with asthma have concurrent atopy (allergic inflammation), which is associated with an improved response to ICS. However, the absence of an atopic phenotype is associated with a poorer ICS response, leaving clinicians with limited treatment options. The nonatopic asthma phenotype has been characterized as the absence of atopic diseases including allergic rhinitis, eczema, or food allergies, and a negative skin prick test to common aeroallergens. Children with mild asthma treated with ICS over 44 weeks without a positive allergen skin test are 3 times more likely to have an asthma exacerbation when compared with children with positive skin tests. Similarly, adolescents and adults with asthma with low blood eosinophils or low sputum eosinophils have no difference in exacerbation rate response to ICS compared with placebo. Due to poor ICS response in nonatopic children and the known adverse effects of ICS, the development of non-steroid treatments options is needed.

Monotherapy with the long-acting muscarinic antagonist, tiotropium, was superior to placebo for treatment failure outcomes in adolescents and adults with low sputum eosinophil levels. Tiotropium is approved in children as an add on therapy to ICS in children ≥ 6 years with asthma. But, this combination of treatment would still expose children with nonatopic asthma to the risks (but potentially without the benefit) of ICS therapy. The objective of this study is to conduct a feasibility pilot safety study of 6-weeks treatment with tiotropium monotherapy vs. ICS in children ages 6 to 11 years old with nonatopic mild persistent asthma.

DETAILED DESCRIPTION:
Asthma Phenotype Variations Suggest the Need for Improved Tailoring of Treatment Options Asthma is the most common chronic disease among children worldwide. Asthma is characterized by chronic airway inflammation; symptoms vary by intensity and frequency over time. The asthma phenotype (observable characteristics such as symptoms and pulmonary function) may present similarly in children, but differences in the underlying endotypes (pathophysiological and/or molecular mechanisms, e.g.T-helper type 2 cell (Th2)-low and Th2-high asthma) indicate that varying processes are present that can affect treatment response Established guidelines (Global Initiative for Asthma [GINA] and National Heart Lung and Blood Institute [NHLBI]) recommend inhaled corticosteroids (ICS) as first line therapy in all children with persistent asthma to manage the inflammatory process and thus, control symptoms (wheeze, shortness of breath, cough, nocturnal awakenings). Yet, currently, 22%-60% of children with asthma continue to present with symptoms or remain poorly controlled while treated according to the established guidelines, which include ICS. Thus, additional studies are needed in children with phenotypes that are poorly responsive to guideline-based therapy with ICS to identify optimal management.

Because asthma phenotypes present similarly (though differing by severity), ICS continue to be the first line of treatment for patients with persistent asthma despite potential differences in underlying pathophysiology (Th2-low and Th2-high endotype). In a controlled trial in children with mild to moderate persistent asthma, 55% were unresponsive to monotherapy treatment with either ICS or montelukast despite over 90% adherence by dose counting. Response to ICS treatment has been associated with several markers of an allergic phenotype that include higher serum eosinophil cationic protein (or serum eosinophil levels), elevated serum IgE, skin test positivity, and elevated exhaled nitric oxide. Indeed, children with mild asthma treated with ICS over 44 weeks who have a positive allergen skin test are 70% less likely to have an asthma exacerbation when compared with children without positivity.

Poor asthma control associated with inadequate treatment response is associated with more health care provider visits, direct costs, and work absenteeism than those with well-controlled asthma. Biomarker-driven asthma management has been suggested as an emerging strategy to improve asthma control by matching treatment selection to underlying endotype (Th2 low vs. Th2 high asthma) differences in pathophysiology. An understudied population of children with asthma are those who lack an allergic phenotype. Treatment response to ICS is poor in this population, but studies have been limited to subgroup analysis from larger populations of mixed phenotypes. Therefore, those children who lack an allergic phenotype may not be optimally treated with guideline-recommended ICS therapy and require studies focused on this phenotype.

Variability in the Definition of the Nonatopic Asthma Phenotype The nonatopic asthma phenotype has been incompletely described and published studies often report varying characteristics. Typical characteristics include the absence of atopic diseases such as allergic rhinitis, eczema, or food allergies; having normal serum IgE levels; and having normal serum eosinophil levels. The most common factor identifying the child with nonatopic asthma is a negative skin prick test (SPT) to common aeroallergens in combination with physician-diagnosed asthma.

Inhaled Corticosteroid Response in Children with Nonatopic Asthma is Suboptimal, and Treatment Options are not Well Studied.

The nonatopic asthma endotype is characterized by a predominantly neutrophilic inflammation of the airway (Th2-low asthma), whereas children with atopic asthma more commonly have elevated airway eosinophils (Th1-high asthma). Numerous studies have found that children with atopic disease (eosinophilic airway inflammation) have a beneficial response to inhaled corticosteroids. However, studies of children with well-characterized non-atopic (predominately neutrophilic versus eosinophilic airway inflammation) are lacking. In large studies to evaluate treatment response of children (~300 participants/trial) with mild to moderate asthma, 20% had negative SPT yet the results of these studies report response rate for the population as a whole, thereby omitting a differential response rate according to atopic status.

Children who do not respond to low doses of ICS (symptoms are not controlled) have therapy augmented with a leukotriene receptor antagonist (montelukast), a long-acting inhaled beta2 agonist, or a higher dose of ICS according to established treatment guidelines. Interestingly, a recent systematic review of 30 trials in children suggests that varying phenotypic characteristics may be useful in identifying children who may respond to a specific class of treatment. In particular, children without a history of eczema regardless of race or ethnicity may have a better response to added bronchodilator treatment (long-acting inhaled beta2 agonist) compared with other treatment choices when combined with ICS therapy. These data are important because it suggests that bronchodilator therapy such as long-acting inhaled beta2 agonist or long-acting muscarinic antagonists (e.g. tiotropium) may have a role as a treatment option in children who lack atopic features.

In the initial treatment of mild persistent asthma for all ages, ICS or montelukast may be used as monotherapy. Treatment with ICS corticosteroids is not without risk in children and has been associated with growth suppression, adrenal suppression, oral candidiasis, and other effects. In addition, these medications can be expensive which potentially contributes to poor adherence. However, montelukast is no longer used as commonly due to modest effects on asthma control and the potential for neuropsychiatric adverse effects. Long-acting inhaled beta2 agonists are not indicated as monotherapy in asthma due to the lack of anti-inflammatory properties but may have synergistic effects when used with an ICS. Long-acting muscarinic antagonists (tiotropium) are currently indicated only for moderate to severe persistent asthma in conjunction with ICS in children 6 years and older. Therefore, new therapeutic options are needed for young children with asthma with mild persistent asthma.

There are no studies which have prospectively examined treatment response in children with nonatopic asthma. A post-hoc analysis that examined biomarkers of response to an ICS (fluticasone) or montelukast in children with mild to moderate asthma, found that those who had lower atopic characteristics (low blood total eosinophil count, low serum eosinophil cationic protein, low serum IgE), and low fraction of exhaled nitric oxide) were less likely to respond to treatment with ICS. In another post-hoc analysis of children with mild asthma treated with inhaled beclomethasone (an ICS), those who lacked skin test positivity or had a lower serum IgE were 70% and 85%, respectively, more likely to experience an exacerbation requiring treatment with ICS.

Evidence of tiotropium effectiveness and safety in patients with asthma and low eosinophilic burden Tiotropium is a long-acting muscarinic antagonist. By blocking the activity of the muscarinic receptor, tiotropium offers an alternative pathway to decrease the airway reactivity, mucus secretion, and inflammation (in vitro). There are recent data to suggest that tiotropium monotherapy is effective and safe in adolescents and adults with mild persistent asthma. Participants with mild persistent asthma were randomized to mometasone (an ICS), tiotropium, or placebo monotherapy in a crossover design with a primary outcome of asthma control. Of those with a low sputum eosinophil level (<2%), 57% had a better response to ICS, and 60% had a better response to tiotropium vs. placebo (essentially no difference between ICS and tiotropium when compared with placebo). Conversely, of those with a high sputum eosinophil level, 74% had a better response to mometasone, and 57% had a better response to tiotropium vs. placebo indicating that Th2-high asthma is preferentially responsive to ICS. Thus, these data confirm that those with a high sputum eosinophil level (greater atopic driven asthma) have a better response to ICS, but the choice between an ICS and tiotropium in those with low sputum eosinophils is less clear. Despite having a low sputum eosinophil level, 80% of participants had at least one positive allergen test at baseline, indicating a component of atopy was still present. In the present pilot study, we will compare the safety of tiotropium monotherapy vs ICS monotherapy in children who have been carefully defined as having mild persistent asthma with a nonatopic phenotype. We expect that the asthma control safety outcomes after treatment with tiotropium will be similar to outcomes after treatment with ICS. Additionally, results from this study may indicate the need to study more effective treatment options for non-atopic asthma.

PRELIMINARY STUDIES/PROGRESS REPORT We have preliminary data from a secondary analysis of the previously described study of ICS and tiotropium in patients with mild persistent asthma (manuscript submitted Blake and Lang, co-authors). We found that in adolescents, the Th2-high biomarkers, aeroallergen positivity (# of positive specific IgE) and ln(IgE) predicts response to ICS [AUC (95% CI), 0.69 (0.52-0.85), p=0.028 and 0.73 (0.58-0.87), p=0.002, respectively]. No Th2-high biomarker data predicts response to tiotropium. However, a phenotypic marker of airway responsiveness (post-albuterol Forced Expiratory Volume in 1 second) did predict response to tiotropium in adolescents (AUC 0.77 0.60-0.95), p=0.002. These data suggest that adolescents without Th2-high asthma (e.g. a nonatopic phenotype) may be less responsive to ICS.

RESEARCH DESIGN AND METHODS INCLUDING STATISTICAL ANALYSIS

Specific Aim and Hypothesis:

Specific Aim 1 is to conduct a randomized crossover pragmatic feasibility pilot safety study of 6-weeks treatment with tiotropium monotherapy vs. ICS in children ages 6 to 11 years old with nonatopic mild persistent asthma. The hypothesis is that there will be no important differences in safety assessments (asthma control, adverse events) between tiotropium and ICS therapy that would preclude moving forward with a larger clinical trial and that evidence of improved asthma control may be observed with tiotropium.

Study Design:

This is a prospective, randomized, open-label crossover pilot feasibility trial. Children with controlled nonatopic mild-persistent asthma ages 6 to 11 years old will be enrolled. Children will be randomized to 6 weeks treatment with tiotropium or ICS followed by a 2-week washout and then randomized to the alternate treatment. This design was used in the trial of tiotropium and ICS in adolescents and adults with asthma described in section Participants will be assessed at 4 visits (baseline, following the 6-week initial treatment period, at the end of the 2-week washout (start of alternative treatment 6-week period), and following alternate 6-week treatment period). Asthma worsening will be assessed in real time using the Daily Digital Diary. Participants will be recruited from the Pulmonology and Allergy Divisions at Nemours Jacksonville. See study schema below. All participants will be provided an Asthma Action Plan at baseline as needed.

Tiotropium and ICS Treatments:

Tiotropium (Spiriva® Respimat®, Boehringer Ingelheim International) is approved as a once-daily maintenance treatment of asthma in patients 6 years and older. The approved dose is 2.5mcg once daily delivered as 2 inhalations of 1.25mcg/inhalation in patients and is typically administered on background treatment with ICS. This dose has been previously studied in children ages 6 to 11 years with moderate to severe asthma. Because we are proposing to use tiotropium as monotherapy, Dr. Vazquez contacted the FDA in December 2020 and an IND submission was recommended.

ICS therapy will be at the drug and dose determined by the treating physician and available through the participant's insurance. ICS will not be provided as part of this trial. Tiotropium is budgeted for this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 6 to 11 years with controlled mild nonatopic persistent physician diagnosed asthma

   1. Non-atopic asthma: absence of a positive SPT to inhaled aeroallergens or negative specific IgE to a common regional allergen panel; historical serum IgE less than 200 IU/ml; historical serum eosinophils less than 350 cells per microliter (cells/mcL); no history of eczema; no history of allergic rhinitis; no history of food allergy
   2. Physician-diagnosed asthma: positive family history, recurrent asthma symptoms, bronchodilator responsiveness, and evidence of obstruction.
   3. Mild persistent asthma: current treatment with as-needed albuterol or low-dose ICS or daily montelukast (Step 2 therapy)
   4. Controlled asthma: Childhood Asthma Control Test score >19
2. Pre-bronchodilator FEV1 ≥ 80% of predicted

Exclusion Criteria:

1. Oral corticosteroid use in the past 6 weeks
2. Use of ICS in combination with long-acting beta agonist or montelukast
3. History of life-threatening asthma requiring treatment with intubation or mechanical ventilation within the past 5 years
4. Respiratory tract infection within the past 4 weeks
5. Any other chronic diseases or medical conditions (other than asthma) that in the opinion of the investigator would prevent participation in a trial

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Change in c-ACT score between standard therapy (inhaled corticosteroids) and tiotropium | The c-ACT will be collected during visit #1 in day 1; visit #2 after 6 weeks at the end of the first arm; visit #3 after 8 weeks at the end of the "wash-out period"; and visit #4 after 14 weeks at the last visit.
  The primary outcome is change in asthma control from baseline to the end of 6-weeks treatment with tiotropium versus ICS. Asthma control will be assessed by the Childhood Asthma Control Test (c-ACT) score. The c-ACT is well validated for assessing asthma control in children aged 4-11 years.41 The c-ACT ranges from 0 to 27; a score of 19 indicates inadequately controlled asthma.

SECONDARY OUTCOMES:
Spirometry FEV1 | The Spirometry FEV1 will be collected during visit #1 in day 1; visit #2 after 6 weeks at the end of the first arm; visit #3 after 8 weeks at the end of the "wash-out period"; and visit #4 after 14
  The National Heart Lung and Blood Institute Guidelines for the Diagnosis and Management of Asthma categorizes lung function measured as the Forced Expiratory Volume in the first second (FEV1) % predicted of normal into three levels: 1) above 80% predicted, typical of mild asthma (both intermittent and persistent); 2) 60% to 80% predicted, typical of moderate persistent asthma; and 3) below 60% predicted, typical of severe persistent asthma. We will compare the change in FEV1 % predicted over the treatment period for tiotropium versus ICS.
Fractional Exhaled Nitric Oxide (FeNO) | The Fractional Exhaled Nitric Oxide (FeNO) will be collecte on day #1 duringf the first visit.
  Biomarker for atopy and will be collected at baseline to be used as covariates in the analysis.
Complete Blood Count with Differential (CBC) | The Complete Blood Count with Differential (CBC) will be collecte on day #1 duringf the first visit.
  Biomarker for atopy and will be collected at baseline to be used as covariates in the analysis.
Daily Digital Diary | The subjects will answer the Daily Digital Diary every day from day 1 until the completion of the study at 14 weeks.
  Asthma symptoms will be assessed using a real-time electronic diary card to capture daily asthma symptoms. This electronic diary card was developed by Dr. Blake for a pilot study funded by the American Lung Association to capture episodes of respiratory tract infections causing respiratory distress in young children. The electronic diary will be modified for this study to capture asthma exacerbations and symptom load. Briefly, each morning, the parent will receive a text with a link to a survey (from REDCap) with a single question "Has your child had had any asthma symptoms in the past 24 hours?" If the parent responds 'yes', a further survey will open to ask albuterol use, prednisone use, unscheduled contact, and frequency of asthma episodes in the past 24 hours that may be an early indication of worsening asthma control.

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo A Vazquez Garcia, MD, Principal Investigator — Nemours
Locations (1):
- Nemours Specialty Care, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided